CLINICAL TRIAL: NCT04707092
Title: Use of Preoperative and Postoperative Antimicrobial Treatment
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 3486
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Ear Infection Bacterial; Surgical Site Infection; Antibiotic Side Effect
MeSH Terms: conditions — Surgical Wound Infection | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Intervention Model Description: Randomization in two treatment arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antibiotic at induction (Experimental): Patients will receive one single dose of Antibiotic at induction
  Interventions: Drug: Antibiotic
- Antibiotic one week (Experimental): Patients will receive one single dose of Antibiotic at induction, plus a 7 day treatment with oral Antibiotic
  Interventions: Drug: Antibiotic

INTERVENTIONS:
Drug: Antibiotic — Antibiotic in case of now allergies will be Cefazolin at induction and Amoxicillin plus Clavulanic acid for the oral treatment week

SUMMARY:
In this study, patients undergoing ear surgery (cochlear implantation, stapedotomy, tympanoplasty) will be randomized to one of two antibiotic treatment groups.

One group will receive a single treatment with an antibiotic at induction

The other group will receive the single intravenous treatment, plus a one week course or oral antibiotic

DETAILED DESCRIPTION:
1. Patients will be asked to participate in the study.
2. Randomization
3. Surgery
4. Follow-up at 1 week, 1 month patients will be asked if they filled their prescription, took the medication as prescribed, experienced any symptoms such as rash, diarrhea, nausea,.. Further the wound will be inspected for any signs of infection. Patients will also be asked if they had noticed discharge, pain, pulsating sensation
5. Follow-up at three months, 1 year and 2 years - patients will again be asked for any signs of infections or necessary visits with their doctor due to infections

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the study
* Undergoing standard ear surgery (Stapedotomy, cochlear implantation, tympanoplasty and tympanomastoidectomy)

Exclusion Criteria:

* multiple allergies to antibiotic substances
* therapy with an antibiotic substance within the last 6 weeks
* prior radiation to the head and neck patients undergoing revision surgery
* Any use of post-operative antibiotics (oral, intravenous, topical) for reason which do not include surgical site infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 1 month
  Side effects from treatment with antibiotics

SECONDARY OUTCOMES:
Infection of surgical site (immediate) | 1 month
  Infection of surgical site with discharge, redness, fever
Infection of surgical site (long term) | 2 years
  infection of surgical site with discharge, fever, extrusion of device

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Center, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No
The individual participant data will not be shared since no conclusions can be drawn from single patient data, the results will be made available in detail